CLINICAL TRIAL: NCT06944353
Title: Improving Diagnostic Safety Through STeatosis Identification, Risk Stratification, and Referral in the ED (STIRRED)
Brief Title: Improving Diagnostic Safety Through STeatosis Identification, Risk Stratification, and Referral in the ED
Acronym: STIRRED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Principal Investigator, Amy Kontrick, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HS029777 (AHRQ); R01HS029777 (AHRQ)
Record Dates: First submitted 2025-04-16; First posted 2025-04-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Steatosis of Liver; Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Metabolic Associated Steatotic Liver Disease; Incidental Radiology finding; Emergency Medicine
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Includes any patient notification about steatosis, education and referrals as per the treating clinician's usual and customary practice.
- STIRRED (Experimental): Patients with incidentally noted hepatic steatosis who are seen in Emergency Departments after STIRRED intervention has been activated within the local EHR may receive additional notification about steatosis, education or referrals for additional testing and follow-up as prompted by the STIRRED intervention which is directed at their discharging clinician.
  Interventions: Behavioral: STIRRED

INTERVENTIONS:
Behavioral: STIRRED — The STIRRED intervention is a behavioral intervention directed at the treating ED clinicians.
  An Our Practice Advisory (OPA) will alert the clinician to the radiology finding of hepatic steatosis at the time of preparing the discharge materials. The OPA will prompt the clinician to discuss this finding with the patient and will automatically add hepatic steatosis to the discharge diagnoses and insert patient-facing discharge information about hepatic steatosis. It will additionally prompt the clinician to refer the patient for follow-up which will be stratified based on their fibrosis risk level.
  Arms: STIRRED

SUMMARY:
Hepatic steatosis is a common radiographic "incidental finding" that is overlooked and underreported to patients. The investigators developed a clinical decision support system using machine learning and natural language processing that will prompt reporting to patients and provide ED clinicians risk stratified follow-up care recommendations. Data on both the implementation and effectiveness of our intervention resulting from this trial will inform future use with a goal of ultimately improving diagnostic safety and outcomes for patients with hepatic steatosis.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is a public health crisis affecting one third of the US adult population. Steatotic liver disease is an obesity related disease with serious health and quality of life consequences. Hepatic steatosis is reported on ~10% of written radiology reports. Unfortunately, lack of awareness often leads to hepatic steatosis being overlooked by providers and unreported to patients leading to delays in diagnosis and referral to specialty care.

This project, Improving Diagnostic Safety through STeatosis Identification, Risk stratification, and Referral pathway in the ED (STIRRED), proposes to improve diagnostic safety by ensuring that patients receive timely notification of the new finding and referral to follow up care. The STIRRED CDSS intervention employs natural language processing and machine learning to identify hepatic steatosis in written emergency department (ED) radiology reports and combine it with common clinical data in the electronic health record to create an individualized risk profile and follow up recommendations for patients with suspected MASLD. This recommendation is communicated to the ED clinician during the ED discharge process via an OurPractice Advisory (OPA) and triggering outpatient referral for follow-up care stratified by risk level.

This trial will evaluate STIRRED across a large health system using a type 2 implementation-effectiveness stepped wedge cluster randomized trial across 11 Emergency Departments in a single health system. Effectiveness of providing risk-based care linkage and implementation outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* imaging finding of hepatic steatosis on ED imaging study
* discharged from the ED to home
* first Northwestern Medicine ED visit in the study period with a hepatic steatosis finding

Exclusion Criteria:

* admitted to the hospital
* age < 18
* pre-existing Liver Disease diagnosis (Liver Cancer, HCV, HBV, Cirrhosis, NAFLD/MASLD/NASH/MASH, Alcohol Liver Disease, PSC, PBC and autoimmune hepatitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4704 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: New steatotic liver disease-related diagnosis among high-risk patients | 120 days post-ED discharge
  For patients at high risk for liver fibrosis, The investigators will evaluate for new steatotic liver disease related ICD codes.
Implementation: Intervention fidelity | Baseline at time of intervention delivery
  Fidelity is the degree to which the STIRRED CDSS was delivered as intended.
  Fidelity will be evaluated across four components:
  1. hepatic steatosis added to the ED discharge diagnoses;
  2. hepatic steatosis patient education provided;
  3. ED adoption of confirming that the clinicians have informed the patient of the new finding; and
  4. ED adoption of placing referral and/or recommendation for follow-up (distinct from routing the message to PCP).
  The Investigators will analyze individual components and a composite score of 0-4 that combines these outcomes. The fidelity components and their composite score (0-4) will be audited monthly from 3 months prior to implementation to 3 months after implementation.

OTHER OUTCOMES:
Effectiveness: New steatotic liver disease-related diagnosis among all patients | 120 days post-ED discharge, 1 year post-ED discharge
  For all patients with incidentally discovered hepatic steatosis, the investigators will evaluate for new steatotic liver disease related ICD codes.
Effectiveness: Non-invasive testing (NIT) completion | 1 year post-ED discharge
  completion of a fibroscan, liver ultrasound, liver elastography, MRI abdomen, MR Elastography or Enhanced Liver Fibrosis(ELF) that indicate ongoing diagnostic process
Effectiveness: new liver lab test completion | 1 year post-ED discharge
  Completion of three key liver disease related lab tests (Liver Function tests, Hepatitis serologies [Hepatitis C Antibody, Hepatitis B surface antigen, Hepatitis B Core antibody, Hepatitis B surface antibody] and INR level) that indicate ongoing diagnostic process;
Effectiveness: new medication initiation | 1 year post-ED discharge
  Receipt of a new prescription for a medication known to impact steatotic liver disease outcomes (e.g., pioglitazone, vitamin E, GLP1 agonist, SGLT2 inhibitor) as an indicator of engagement in lifestyle changes and weight loss interventions.
Effectiveness: new referrals | 1 year post-ED discharge
  Receipt of referral to lifestyle medicine (nutrition) or bariatric surgery as an indicator of engagement in lifestyle changes and weight loss interventions.
Effectiveness: weight change | 1 year post-ED discharge
  Weight values for patients will be evaluated when available to assess for weight loss over time as an indicator of engagement in lifestyle changes and weight loss interventions.
Implementation: Acceptability of Intervention Measure (AIM) | 2 months after STIRRED implementation; 4 months after final site STIRRED implementation
  Acceptability is the perception that STIRRED is satisfactory or agreeable to ED clinicians
Implementation: Intervention Appropriateness Measure (IAM) | 2 months after STIRRED implementation; 4 months after final site STIRRED implementation
  Appropriateness is the perceived fit or compatibility of STIRRED for the ED and ED patients
Implementation: Feasibility of Intervention Measure (FIM) | 2 months after STIRRED implementation; 4 months after final site STIRRED implementation
  feasibility is the extent to which STIRRED can be used within the course of an ED clinical encounter
Implementation: Clinical Sustainability | 2 months after STIRRED implementation; 4 months after final site STIRRED implementation
  The Clinical Sustainability Assessment Tool (CSAT) will be used to understand factors that contribute to sustainability of the STIRRED model in practice over time from the perspective of the ED clinicians.
Implementation: Cognitive Load of Intervention | 2 months after STIRRED implementation; 4 months after final site STIRRED implementation
  NASA task load index (TLX) will assess cognitive load of STIRRED for the ED clinicians. The NASA TLX is a 6-item instrument that has been used to measure the workload of a system.

CONTACTS AND LOCATIONS:
Overall Officials: Amy V Kontrick, MD, Principal Investigator — Northwestern University; Danielle M McCarthy, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD used in the analysis of the hybrid implementation effectiveness trial will be shared. All published data will be formatted according to the principals of Common Data Elements (CDE) as defined by the NIH. Clinical and survey response data will contain raw item responses as well as any aggregate scores for participants. To facilitate future use and interoperability of our data, we will employ standard processing and documentation protocols adopted by the Inter-university Consortium for Political and Social Research (ICPSR) for data formats and dictionaries as well as for variable names, descriptions, and labels.
  Data will be made available through a data repository (still to be determined) following the completion of the grant period and final publication of the trial manuscript.

REFERENCES:
- [Derived] McCarthy DM, VanWagner LB, Rafferty MR, Cameron KA, Lee J, Dong S, Fellner A, Kontrick AV. Improving diagnostic safety through steatosis identification, risk stratification, and referral pathway in the ED (STIRRED): Protocol for an effectiveness implementation trial. Contemp Clin Trials. 2025 Dec 15;161:108187. doi: 10.1016/j.cct.2025.108187. Online ahead of print. PMID 41407098